CLINICAL TRIAL: NCT05258110
Title: The Effect of Multiple Oral Doses of BI 425809 on Metabolism of Midazolam Administered Orally in Healthy Male Subjects (Open-label, Two-period, One-sequence Trial)
Brief Title: A Study in Healthy Men to Test Whether BI 425809 Influences the Amount of Midazolam in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0035; 2021-005585-17 (EudraCT Number)
Record Dates: First submitted 2022-02-24; First posted 2022-02-28 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Solutions; BI 425809

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference (R): midazolam alone (Experimental): First treatment period
  Interventions: Drug: midazolam
- Test (T): midazolam + BI 425809 (Experimental): Second treatment period
  Interventions: Drug: midazolam; Drug: BI 425809

INTERVENTIONS:
Drug: midazolam — midazolam
  Other Names: Midazolam-ratiopharm® 2 mg/ml solution
Drug: BI 425809 — BI 425809
  Arms: Test (T): midazolam + BI 425809

SUMMARY:
In order to assess the potential impact of steady state BI 425809 on CYP3A clinically, the effect of BI 425809 on the midazolam pharmacokinetics will be evaluated. Midazolam is a recommended substrate of CYP3A4.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 millimetre of mercury (mmHg), or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of midazolam in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 12 hours per each period
Maximum measured concentration of midazolam in plasma (Cmax) | up to 12 hours per each period

SECONDARY OUTCOMES:
Area under the concentration-time curve of midazolam in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 12 hours per each period

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com